CLINICAL TRIAL: NCT00368680
Title: Early Bubble CPAP (EBCPAP) in Very Low Birth Weight Infants (VLBWI)
Brief Title: Early CPAP in Respiratory Distress Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Neonatologia, Hospital Clinico, Pontificia Universidad Catolica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEO032006
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2007-04

CONDITIONS: Respiratory Distress Syndrome
Keywords: Respiratory Distress Syndrome; Early Bubble CPAP; Mechanical Ventilation; Surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome

INTERVENTIONS:
Device: Early Bubble CPAP

SUMMARY:
The purpose of this study is to establish if a strategy of EBCPAP application in a subgroup of VLBWI, 800 to 1500g birthweight, decreases the need for mechanical ventilation in this group, without affecting mortality.

DETAILED DESCRIPTION:
The application of CPAP has been described as an alternative respiratory support for premature newborns with respiratory distress.Many studies support that the early use of CPAP results in a better respiratory evolution and less need for mechanical ventilation.

Hypothesis:

- The hypothesis is that EBCPAP will decrease the need for this more invasive therapy.

The primary endpoint in this multicenter controlled study is to establish if an strategy of EBCPAP application in a subgroup of VLBWI, 800 to 1500g birthweight, decreases the need for mechanical ventilation in this group, without affecting mortality. .

As secondary outcome, the investigators will analyse: days of oxygen therapy, days of mechanical ventilation, need for surfactant , pulmonary airleak, intraventricular hemorrhage, persistent ductus arteriosus, retinopathy of prematurity and bronchopulmonary dysplasia (BPD) at 28 days and 36 weeks corrected gestational age.

Comparison(s):

Early Bubble CPAP (EBCPAP)with Standard Therapy which is oxygen.

ELIGIBILITY:
Inclusion Criteria:

* All infants born at the units belonging to the South American Neocosur Network with a birthweight between 800 to 1500g and breathing spontaneously at birth or after hand bagging with Neopuff or transient intubation are eligible.
* An informed consent form should be obtained preferable prenatal.

Exclusion Criteria:

* Acute life threatening congenital malformations or genetics diseases.
* Apgar score equal or less than 3 at 5 minutes
* Disapproval of informed consent.

Ages: 5 Minutes to 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-04; Study Completion 2009-09

PRIMARY OUTCOMES:
Need for mechanical ventilation

SECONDARY OUTCOMES:
Days of oxygen therapy
Days of mechanical ventilation
Need for surfactant
Pulmonary airleak
Intraventricular hemorrhage
Persistent ductus arteriosus
retinopathy of prematurity
Bronchopulmonary dysplasia (BPD) at 28 days and 36 weeks corrected gestational age.

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Tapia, MD, Principal Investigator — Pontificia Universidad Católica; Aldo Bancalari, MD, Principal Investigator — Hospital Guillermo Grant; Soledad Urzua, MD, Principal Investigator — Pontificia Universidad Católica
Locations (14):
- Argentina (5):
  - Servicio de Neonatología, Hospital de Clínicas José de San Martín, Buenos Aires
  - Servicio de Neonatología, Hospital Fernández, Buenos Aires
  - Servicio de Neonatología, Hospital Italiano, Buenos Aires
  - Servicio de Neonatología, Maternidad Sardá, Buenos Aires
  - Servicio de Neonatología, Hospital Lagomaggiore, Mendoza
- Chile (6):
  - Servicio de Neonatología, Hospital Gustavo Fricke, Viña del Mar, Región de Valparaíso
  - Servicio de Neonatología, Hospital Guillermo Grant, Concepción, Región del Biobío
  - Servicio de Neonatología, Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan
  - Servicio de Neonatología, Hospital San José, Santiago, Santiago Metropolitan
  - Servicio de Neonatología, Hospital Sótero del Rio, Santiago, Santiago Metropolitan
  - Unidad de Neonatología, Hospital Clínico Pontificia Universidad Católica, Santiago, Santiago Metropolitan
- Servicio de Neonatología, Hospital de Clinicas Universidad Nacional Asunción, Asunción, Paraguay
- Servicio de Neonatología, Hospital Cayetano Heredia, Lima, Peru
- Servicio de neonatología, Centro Hospitalario Pereira Rosseli, Montevideo, Uruguay

REFERENCES:
- [Background] Gregory GA, Kitterman JA, Phibbs RH, Tooley WH, Hamilton WK. Treatment of the idiopathic respiratory-distress syndrome with continuous positive airway pressure. N Engl J Med. 1971 Jun 17;284(24):1333-40. doi: 10.1056/NEJM197106172842401. No abstract available. PMID 4930602
- [Background] Krouskop RW, Brown EG, Sweet AY. The early use of continuous positive airway pressure in the treatment of idiopathic respiratory distress syndrome. J Pediatr. 1975 Aug;87(2):263-7. doi: 10.1016/s0022-3476(75)80599-3. PMID 1097619
- [Background] Allen LP, Reynolds ER, Rivers RP, Le Souef PM, Wimberley PD. Controlled trial of continuous positive airway pressure given by face mask for hyaline membrane disease. Arch Dis Child. 1977 May;52(5):373-8. doi: 10.1136/adc.52.5.373. PMID 326199
- [Background] Hegyi T, Hiatt IM. The effect of continuous positive airway pressure on the course of respiratory distress syndrome: the benefits on early initiation. Crit Care Med. 1981 Jan;9(1):38-41. doi: 10.1097/00003246-198101000-00009. PMID 6780266
- [Background] Kamper J, Wulff K, Larsen C, Lindequist S. Early treatment with nasal continuous positive airway pressure in very low-birth-weight infants. Acta Paediatr. 1993 Feb;82(2):193-7. doi: 10.1111/j.1651-2227.1993.tb12637.x. PMID 8477167
- [Background] Kamper J. Early nasal continuous positive airway pressure and minimal handling in the treatment of very-low-birth-weight infants. Biol Neonate. 1999 Jun;76 Suppl 1:22-8. doi: 10.1159/000047043. PMID 10393390
- [Background] Lundstrom KE. Initial treatment of preterm infants--continuous positive airway pressure or ventilation? Eur J Pediatr. 1996 Aug;155 Suppl 2:S25-9. doi: 10.1007/BF01958077. PMID 8839743
- [Background] Van Marter LJ, Allred EN, Pagano M, Sanocka U, Parad R, Moore M, Susser M, Paneth N, Leviton A. Do clinical markers of barotrauma and oxygen toxicity explain interhospital variation in rates of chronic lung disease? The Neonatology Committee for the Developmental Network. Pediatrics. 2000 Jun;105(6):1194-201. doi: 10.1542/peds.105.6.1194. PMID 10835057
- [Background] Michna J, Jobe AH, Ikegami M. Positive end-expiratory pressure preserves surfactant function in preterm lambs. Am J Respir Crit Care Med. 1999 Aug;160(2):634-9. doi: 10.1164/ajrccm.160.2.9902016. PMID 10430740
- [Background] Verder H, Albertsen P, Ebbesen F, Greisen G, Robertson B, Bertelsen A, Agertoft L, Djernes B, Nathan E, Reinholdt J. Nasal continuous positive airway pressure and early surfactant therapy for respiratory distress syndrome in newborns of less than 30 weeks' gestation. Pediatrics. 1999 Feb;103(2):E24. doi: 10.1542/peds.103.2.e24. PMID 9925870
- [Background] Ho JJ, Henderson-Smart DJ, Davis PG. Early versus delayed initiation of continuous distending pressure for respiratory distress syndrome in preterm infants. Cochrane Database Syst Rev. 2002;2002(2):CD002975. doi: 10.1002/14651858.CD002975. PMID 12076463
- [Background] Subramaniam P, Henderson-Smart DJ, Davis PG. Prophylactic nasal continuous positive airways pressure for preventing morbidity and mortality in very preterm infants. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD001243. doi: 10.1002/14651858.CD001243.pub2. PMID 16034858
- [Background] Lee KS, Dunn MS, Fenwick M, Shennan AT. A comparison of underwater bubble continuous positive airway pressure with ventilator-derived continuous positive airway pressure in premature neonates ready for extubation. Biol Neonate. 1998;73(2):69-75. doi: 10.1159/000013962. PMID 9483299
- [Background] De Klerk AM, De Klerk RK. Nasal continuous positive airway pressure and outcomes of preterm infants. J Paediatr Child Health. 2001 Apr;37(2):161-7. doi: 10.1046/j.1440-1754.2001.00624.x. PMID 11328472
- [Background] Narendran V, Donovan EF, Hoath SB, Akinbi HT, Steichen JJ, Jobe AH. Early bubble CPAP and outcomes in ELBW preterm infants. J Perinatol. 2003 Apr-May;23(3):195-9. doi: 10.1038/sj.jp.7210904. PMID 12732855
- [Derived] Tapia JL, Urzua S, Bancalari A, Meritano J, Torres G, Fabres J, Toro CA, Rivera F, Cespedes E, Burgos JF, Mariani G, Roldan L, Silvera F, Gonzalez A, Dominguez A; South American Neocosur Network. Randomized trial of early bubble continuous positive airway pressure for very low birth weight infants. J Pediatr. 2012 Jul;161(1):75-80.e1. doi: 10.1016/j.jpeds.2011.12.054. Epub 2012 Mar 6. PMID 22402568